CLINICAL TRIAL: NCT03765333
Title: Descriptive Observational Epidemiological Study on the Characteristics of Thyroid Cancer in Patients Treated in Oncology Services of Spanish Centers: National Registry of Thyroid Cancer - Differentiated, Medullary and Anaplastic
Brief Title: GETNE Registration of Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Other Study IDs: REGETNE-Tiroides
Record Dates: First submitted 2018-11-20; First posted 2018-12-05 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Thyroid Cancer
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
An epidemiological, observational, multicenter, cross-sectional, retrospective study on patients ≥ 18 years visited in the oncology services of the participating centers with diagnosis of primary thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with diagnosis of differentiated, medullary or anaplastic thyroid cancer confirmed by histopathology.
* Patients who agree to participate and are able to understand the information sheet and sign the informed consent

Exclusion Criteria:

* Patients under 18 years of age.
* Patients with other types of thyroid cancer or whose histopathological diagnosis has not been confirmed.
* Patients who do not have the relevant basic information to be included in the study, according to the criteria of the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥ 18 years visited in the oncology services of the participating centers that have a diagnosis of primary cancer located in the thyroid gland.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hystopathological characteristics of the tumor | Baseline
  Based on pathologist evaluation of biopsy including differentiated, medullar or anaplasic.
Situation of the tumor at first-diagnosis | Baseline
  Local tumor, locoregional tumor or metastatic disease.
Tumor-Node-Metastasis classification | Baseline
  Based on the AJCC (American Joint Committee on Cancer) 2018 TNM system: T for extent or size of the tumor, N for lymph nodes spread and M for metastasis.
Tumor Stage | Baseline
  From I to IV, based on the interpretation of the TNM classification and depending on the hystopathological characteristics of the tumor.

SECONDARY OUTCOMES:
Patient situation at the end of treatment | 12 months
  Results of clinical evaluation of the disease including complete response, partial response, stable disease, progression of disease or death
Number of patients with BRAF mutation | 12 months
  Total patients with available results on BRAF status and proportion of patients with mutated BRAF or native BRAF.
Number of patients with RET mutation | 12 months
  Total patients with available results on RET status and proportion of patients with mutated RET or native RET.
Number of patients with PI3K mutation | 12 months
  Total patients with available results on PI3K status and proportion of patients with mutated PI3K or native PI3K.
Number of patients with RAS mutation | 12 months
  Total patients with available results on RAS status and proportion of patients with mutated RAS or native RAS.
Number of patients with PAX8/PAR mutation | 12 months
  Total patients with available results on PAX8/PAR status and proportion of patients with mutated PAX8/PAR or native PAX8/PAR.
Number of patients with P53 mutation | 12 months
  Total patients with available results on P53 status and proportion of patients with mutated P53 or native P53.
Number of patients with PTEN mutation | 12 months
  Total patients with available results on PTEN status and proportion of patients with mutated PTEN or native PTEN.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Hernando Cubero, M.D., Study Director — Hospital Universitari Vall d'Hebron, Barcelona; Jaume Capdevila, M.D., Study Chair — Hospital Universitari Vall d'Hebron, Barcelona
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No